CLINICAL TRIAL: NCT06253273
Title: Functional Assessment of the Patient With Fibromyalgia and Its Relation to Health: Fibromyalgia and Sarcopenia
Acronym: FIBYSAR
Status: Completed | Type: Observational
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Other Study IDs: CamiloJcUFYS
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia; Sarcopenia
MeSH Terms: conditions — Fibromyalgia; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fibromyalgia is a chronic syndrome that causes fatigue, sleep disorders and generalized chronic pain in different parts of the body. This pathology is more prevalent in women and is generally not attributed to any specific cause.

This observational study aims to describe some important and health-related factors in patients with fibromyalgia.

Participants will have to fill out questionnaires related to sleep, anxiety, impact of the disease and sarcopenia index, and will then take tests related to grip strength for the upper limbs and dynamometry in the lower limbs. We will also employ the use of ultrasound to evaluate architectural measurements. Last but not least, we cannot forget the pain measurements that are so necessary in this study population.

DETAILED DESCRIPTION:
Through the present research study we intend to analyze not only the health status of our sample but also to correlate the parameters analyzed with factors related to sarcopenia.

Through the data collection that will be carried out we can analyze variables as essential as pain, anxiety and depression, impact of the disease, agility, strength, anthropometric measurements, sleep and muscular architectural measurements by means of ultrasound in which we can analyze the fatty infiltration of structures such as the vastus lateralis, rectus anterior and vastus medius that allow us to obtain data that can define the characteristics of patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FM
* aged between 18 and 75 years
* agree to participate and sign the informed consent.

Exclusion Criteria:

* who do not have recent surgeries
* patients with reduced mobility
* adequate level of comprehension to be able to answer the questionnaires that will be provided in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia belonging to the Asocación Afinsyfacro de Móstoles. All men and women of the Association who meet the inclusion and exclusion criteria may participate.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-05-03 (Actual)

PRIMARY OUTCOMES:
Algometer | baseline
  Algometer points: Using an algometer, the pain threshold at each tender point is measured in kg/cm. The higher the value obtained, the less pain the subject has.
VAS | baseline
  Visual Analogic Scale: this self-referenced scale ranges from 0 to 10 where 0 is no pain at all and 10 indicates the worst possible pain endured. The higher the score, the greater the pain
Circometry | baseline
  Contour measurements: The contour of the segment selected for the study will be measured using a tape measure. It is measured in centimeters. the greater the number of centimeters, the greater the diameter and therefore the worse the condition or greater the liquid retention of the subject.
Dynamometer | baseline
  upper limb grip strength: this measuring tool measures upper limb grip strength. the higher the value, the better the subject's state of strength
Iso-pull | baseline
  lower limb strength: this measuring tool measures the strength of lower limbs. the higher the value, the better the subject's state of strength.
Chair test | baseline
  number of squats for 30 seconds: this test consists of seeing how many squats can be done in the test time. The greater the number of squats, the better the subject will be.
Timed up and go | baseline
  balance test: The Timed Up and Go Test is an easy-to-use test to assess the risk of falls.The shorter the test time, the lower the risk of falling.
anthropometric measurements | baseline
  anthropometric measurements with the uso of the Tanita
muscular architectural stockings | baseline
  taking architectural muscle averages using an ultrasound scanner
Pittsburgh | baseline
  sleep quality questionnaire: This test has values from 0 to 21 points maximum. It is interpreted that the higher the score, the worse the quality of sleep.
FIQ | baseline
  fibromyalgia impact questionnaire: The total FIQ score is between 0-100 as each of the items has a score of 0-10 once adapted. Thus, 0 represents the highest functional capacity and quality of life and 100 the worst state.
SARC-F | baseline
  questionnaire to measure sarcopenia risk: The SARC-F is a quick and easy instrument for detecting the risk of sarcopenia, which asks the degree of difficulty an older adult has in performing 4 functional activities. A score greater than 4 indicates risk of sarcopenia.
HADS | baseline
  to evaluate emotional distress in patients with different chronic conditions, assessing cognitive and behavioral symptoms of anxiety and depression. The HADS is composed of two subscales: Depression and Anxiety, each with seven items. The score of each subscale can vary between 0 and 21, since each item presents four response options, ranging from absence/minimal presence = 0, to maximum presence = 3.

SECONDARY OUTCOMES:
socio-demographic variables | baseline
  socio-demographic variables (age, weight, height, medication intake, marital status, employment status, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Úbeda D'ocasar, Principal Investigator — Associate Professor
Locations (1):
- University Camilo José Cela, Madrid, Spain